CLINICAL TRIAL: NCT03345511
Title: Ultrasound Guided Analgesic Caudal Block in Anal Canal Surgery
Brief Title: Ultrasound Guided Caudal Block for Benign Anal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UdeA1001
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2017-02

CONDITIONS: Anal Fissure; Anal Fistula; Hemorrhoids; Pain, Postoperative
Keywords: ultrasound guided caudal block; anal surgery
MeSH Terms: conditions — Fissure in Ano; Rectal Fistula; Hemorrhoids; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound Guided Caudal Block (Experimental): 30 minutes before benign canal anal surgery, a 18 G tuohy needle guided with an ultrasound probe to visualize the caudal space, a solution of bupivacaine 0.25%, Lidocaine 1% and dexamethasone 8mg was injected and needle removed.
  Interventions: Procedure: Ultrasound Guided Caudal Block

INTERVENTIONS:
Procedure: Ultrasound Guided Caudal Block — Using an external ultrasound probe, the investigators guided a 18 gauge epidural needle into the caudal space and injected a local anesthetic solution consisting in bupivacaine 0.25%, lidocaine 1% and dexamethasone 8mg in the caudal space.

SUMMARY:
Interventional study that evaluate analgesia and side effects of Ultrasound guided Caudal block preoperatively in benign canal anal surgery

DETAILED DESCRIPTION:
Postoperative pain is an important symptom in patients after benign anal canal surgery. Caudal block has been described to decrease postoperative pain in this type of surgery. Ultrasound is a tool that facilitates its performance and increases the rate of a successful block.

Objective:

To determine the usefulness of ultrasound guided caudal block in anesthesia and postoperative analgesia in patients scheduled for benign anal surgery. Methods : Interventional study in adult patients that received ultrasound caudal anesthetic block before benign anal surgery. The investigators evaluated analgesic efficacy of this intervention by mean of numeric rating scale ( NRS) for pain after 6, 12 and 24 hours of surgery, rescue analgesia, motor block, urinary retention, surgical conditions and patient satisfaction in postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 70 year old patient
* schedule for benign anal surgery ( hemorrhoids, anal fistula, fissure or abcess )
* Caudal analgesic injection before surgery
* Use of ultrasound to guide needle insertion into caudal space

Exclusion Criteria:

* cognitive impairment
* verbal communication impairment
* infection in skin at injection site
* coagulopathy
* technique refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity (P3). Self reported pain intensity at 6, 12 and 24 hours after surgery. | 1 day
  The pain numeric Rating Scale (NRS) is a single 11-point numeric scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain , with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable")

SECONDARY OUTCOMES:
Rescue Analgesia (R3) need of opioid medication for rescue severe postoperative pain at 6, 12 and 24 hours after surgery. | 1 day
  Doses of intravenous tramadol for rescue in severe postoperative pain

OTHER OUTCOMES:
motor block | 2 hours post surgical
  presence or absence of motor block in lower extremity after caudal block

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Cadavid, MD, Principal Investigator — Anesthesiology Professor
Locations (1):
- hospital universitario San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
only final results of research

REFERENCES:
- [Background] Shin S, Kim JY, Kim WO, Kim SH, Kil HK. Ultrasound visibility of spinal structures and local anesthetic spread in children undergoing caudal block. Ultrasound Med Biol. 2014 Nov;40(11):2630-6. doi: 10.1016/j.ultrasmedbio.2014.06.020. Epub 2014 Sep 12. PMID 25220270
- [Background] Ibacache ME, Munoz HR, Fuentes R, Cortinez LI. Dexmedetomidine-ketamine combination and caudal block for superficial lower abdominal and genital surgery in children. Paediatr Anaesth. 2015 May;25(5):499-505. doi: 10.1111/pan.12642. Epub 2015 Mar 4. PMID 25736098
- [Background] Doo AR, Kim JW, Lee JH, Han YJ, Son JS. A Comparison of Two Techniques for Ultrasound-guided Caudal Injection: The Influence of the Depth of the Inserted Needle on Caudal Block. Korean J Pain. 2015 Apr;28(2):122-8. doi: 10.3344/kjp.2015.28.2.122. Epub 2015 Apr 1. PMID 25852834